CLINICAL TRIAL: NCT02619370
Title: Evaluation of an Advance Care Planning Activity: Feasibility Testing for a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lauren Van Scoy (Other)
Collaborators: University of Kentucky (Other); Francis Family Foundation (Other); Penn State University (Other)
Responsible Party: Sponsor-Investigator, Lauren Van Scoy, Assistant Professor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00002634
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Chronic Disease; Caregivers
Keywords: advance care planning; advance directive; caregiving
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Play 'My Gift of Grace,' a conversation card game for 4-6 players (the game consists of 20 question cards that prompt players to identify and articulate their values and beliefs related to dying and end-of-life issues); all game sessions will be audio recorded and transcribed.
  Interventions: Behavioral: Conversation card game
- Control (Active Comparator): Review and discuss a brochure on ACP called "Advance Care Planning: Tips from the National Institute of Aging". Discussion will be prompted by the researcher asking participants to discuss the information they've just read with the group. However, there will not be a formal structure to this discussion.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Conversation card game
  Arms: Intervention
Behavioral: Active Control
  Arms: Control

SUMMARY:
The overarching goal of this project is to facilitate engagement of individuals in effective advance care planning (ACP). Our specific objective is to conduct a randomized, controlled trial to determine whether playing a structured conversation game will increase the likelihood that participants will complete advance directives and perform other ACP behaviors compared to those who are provided with only standard ACP educational materials.

DETAILED DESCRIPTION:
Our central hypothesis is that having ACP conversations in a non-threatening and enjoyable game format will stimulate participants to engage in additional ACP behaviors including completion of ADs. We will use the ACP Engagement Survey to measure readiness to perform ACP, which includes measures of the "stage of change" for performing ACP behaviors.

The proposed study has two specific aims:

Aim 1. To determine whether individuals who play a conversation game are more likely to subsequently complete an online AD (called 'Making Your Wishes Known'; MYWK) compared to individuals who receive standard information about ACP. Our hypothesis is that playing a conversation game will result in a higher AD completion rate (compared to control) in the three months following the intervention.

Aim 2. To identify which participant and/or conversation-related factors influence movement along the stages of change continuum with respect to ACP behaviors (discussing end-of-life wishes with families or clinicians and then completing ADs). Our hypotheses are that: H1) the game intervention will lead to higher quality conversations than the control; and H2) participants whose conversations consist of high-quality ACP discussions will be more likely to progress toward enacting ACP behaviors (as measured by the ACP Engagement Survey score) than those participants whose conversations consist of low-quality discussions.

ELIGIBILITY:
Participants are eligible to participate if they fall into at least one of the following three groups:

* Group 1) CAREGIVERS:

  * are 18 years or older
  * speak and read English
  * have been an unpaid caregiver for an adult over the age of 18 in the last 12 months. Being an unpaid caregiver may include helping with personal needs or household chores, managing a person's finances, arranging for outside services, or visiting regularly to see how they are doing. This person need not live with participants in order for them to identify as caregivers;
  * are able to sit for about 2.5-3 hours
  * are able to focus on the game for about 1.5-2 hours
  * can complete required survey
  * care recipient is capable of discussing medical issues
  * care recipient has not completed an AD in past 18 months
* Group 2) PATIENTS WITH CHRONIC ILLNESS; criteria include:

  * are 18 years or older
  * speak and read English
  * have at least one chronic illness (cancer, chronic pulmonary disease, coronary artery disease, congestive heart failure, peripheral vascular disease, severe chronic liver disease, diabetes with end organ damage, renal failure-defined using Iezonnis' ICD-9 criteria*)
  * have not completed an advance directive within the past 18 months
  * are able to sit for about 2.5-3 hours
  * are able to focus on the game for about 1.5-2 hours
  * can complete required surveys
* Group 3) SURROGATE DECISION MAKERS FOR PATIENTS WITH CHRONIC ILLNESS criteria include:

  * considers themselves a surrogate decision maker for an adult with a chronic illness (defined by Iezonni's ICD-9 chronic illness categories*)
  * are 18 years or older
  * speak and read English
  * are able to sit for about 2.5-3 hours
  * are able to focus on the game for about 1.5-2 hours
  * can complete required surveys
* Iezonni's ICD-9 'chronic illness' definition contains codes within any of the following categories:

  1. malignant cancer/leukemia
  2. chronic pulmonary disease
  3. coronary artery disease
  4. congestive heart failure
  5. peripheral vascular disease
  6. severe chronic liver disease
  7. diabetes with end-organ damage
  8. renal failure.

Exclusion Criteria:

* Do not fall into one of the above 3 categories
* Are <18 years of age
* Non-English speaking
* Cognitively impaired by self-report or score less than 21 on the MoCA screening tool
* Do not have a chronic illness (lacking one of the diseases from Iezonni's ICD-9 codes in chronic illness categories, described above)
* Have completed an advance directive within the last 18 months
* Do not provide informed consent or unable to provide informed consent
* Carry a diagnosis of dementia
* Unable to complete a 3 hour study session in one sitting (by self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Completion of an online advance directive | 3 months

SECONDARY OUTCOMES:
Advance Care Planning Engagement Survey | 3 months
  This survey includes information about stage of readiness to perform advance care planning, self-efficacy, and other measures of behavioral change
Advance Care Planning Behaviors | 3 months
  Open-ended interviews will ascertain additional advance care planning behaviors performed

OTHER OUTCOMES:
Satisfaction with advance care planning questionnaire | 30 minutes after intervention
  8-item questionnaire on a 7-point likert scale